CLINICAL TRIAL: NCT07402018
Title: Arterial Compliance as a Predictor of Clinical Outcomes With Intra-aortic Balloon Counterpulsation: A Prospective Observational Pilot Study
Brief Title: Intra-aortic Balloon Counterpulsation (IABC) Compliance
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Matthew Delfiner, Principal Investigator: Matthew S Delfiner DO, MS, Thomas Jefferson University
Other Study IDs: 2025-0678
Record Dates: First submitted 2026-01-09; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Cardiogenic Shock; IABC Procedure; Intraaortic Balloon Counterpulsation (IABC)
Keywords: Cardiogenic shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators intend to study how baseline arterial compliance (as defined by stroke volume/pulse pressure) influences the clinical success of intraaortic balloon counterpulsation (IABC) in patients with cardiogenic shock (CS). The investigators aim to compare clinical outcomes in CS patients requiring IABC with normal compliance versus low compliance. The study will enroll patients undergoing IABC that are clinically indicated. Baseline hemodynamic measurements will be obtained and then patients would be stratified based on their compliance. Post IABC, serial hemodynamic measurements will be obtained and compared between groups. Patients will continue to be followed longitudinally until the IABC has been discontinued for any reason. The proposed study will yield results that will aid in developing a larger clinical trial and ultimately assist clinicians in determining if IABC is appropriate therapy for patients in cardiogenic shock.

DETAILED DESCRIPTION:
This study will focus on patients in cardiogenic shock (CS) that will be undergoing clinically indicated intraaortic balloon counterpulsation (IABC) insertion and right heart catheterization. Prior to IABC insertion a patient will have their clinically indicated right heart catheterization. The investigators will record these baseline hemodynamic parameters, including (but not limited to) stroke volume and arterial pulse pressure.

After IABC insertion is completed, repeat hemodynamic measurements will be obtained approximately 30 minutes later. Repeat hemodynamic measurements will be recorded at approximately 3-6 hours following the procedure, and 24 hours following the procedure. The act of recording hemodynamic measurements is part of the usual clinical management of patients with IABC.

The patients will continue be followed longitudinally until their IABC course has completed, either due to resolution of CS, exchange for a separate device, heart transplantation, durable Left Ventricular Assist Device (LVAD) implant, or patient death.

The investigators hypothesize that patients with low arterial compliance will have greater improvements in cardiac output and cardiac filling pressures compared to patients with normal compliance. The specific aims are to (1) compare hemodynamic changes with IABC in cardiogenic shock patients with low compliance vs those with normal compliance and (2) to determine a cutoff value of compliance that can be used for future larger clinical trials.

The proposed study will yield results that will aid in developing a larger clinical trial and ultimately assist clinicians in determining if IABC is appropriate therapy for patients in cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Cardiogenic shock
* Undergoing Intra-aortic Balloon Counterpulsation (IABC) as part of clinical care
* Able to provide consent or have power of attorney or next of kin provide consent

Exclusion Criteria:

* Age <18 years old
* Unable to consent or does not have power of attorney or next of kin to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiogenic shock patients undergoing Intra-aortic Balloon Counterpulsation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output (L/min) | 24 hours

SECONDARY OUTCOMES:
Systolic Blood Pressure (mmHg) | 30 minutes
Pulmonary Artery Oxygen Saturation (%) | 24 hours
Ultimate Disposition | Longitudinal Follow-Up (approximately 3 months)
  Hospital death
Total Bilirubin (mg/dL) | 24 hours
  participant laboratory value
ALT (U/L) | 24 hours
  participant laboratory value
AST (U/L) | 24 hours
  participant laboratory value
Creatine Clearance/GFR | 24 hours
Creatine (mg/dL) | 24 hours
  participant laboratory value
Lactate millimoles per liter (mmol/L) | 24 hours
  participant laboratory value
Pulmonary Artery Compliance (mmHg) | 24 hours
Right Ventricular Stroke Work Index (g·m-²·beat-¹) | 24 hours
Pulmonary Artery Pulsatility Index (PAPi) | 24 hours
  calculated measurement
Pulmonary Vascular Resistance (dynes/cm⁵) | 24 hours
Systemic Vascular Resistance (mmHg/L/min) | 24 hours
Pulmonary Capillary Wedge Pressure (mmHg) | 24 hours
Diastolic Pulmonary Arterial Pressure (mmHg) | 24 hours
Systolic Pulmonary Artery Pressure (mmHg) | 24 hours
Right Atrium Pressure (mmHg) | 24 hours
  report measurement
Aortic Pulsatility Index (API) | 24 hours
  calculated measurement
Cardiac Power Input (W/m²) | 24 hours
Cardiac Power Output (Watts) | 24 hours
Stroke Volume (mL) | 24 hours
Cardiac Index (L/min/m²) | 24 hours
Heart Rhythm | 24 hours
  Normal Sinus Rhythm, Atrial Fibrillation, Atrial Flutter, Ventricular Fibrillation, Ventricular Tachycardia, Sinus Bradycardia, Sinus Tachycardia, other
Heart Rate (beats per minute) | 24 hours
Mean Arterial Pressure (mmHg) | 24 hours
Diastolic Blood Pressure (mmHg) | 24 hours
Systolic Blood Pressure (mmHg) | 24 hours
Pulmonary Artery Compliance (mmHg) | 3-6 hours
Right Ventricular Stroke Work Index (g·m-²·beat-¹) | 3-6 hours
Pulmonary Artery Pulsatility Index (PAPi) | 3-6 hours
  calculated measurement
Pulmonary Vascular Resistance (dynes/cm⁵) | 3-6 hours
Systemic Vascular Resistance (mmHg/L/min) | 3-6 hours
Pulmonary Capillary Wedge Pressure (mmHg) | 3-6 hours
Diastolic Pulmonary Arterial Pressure (mmHg) | 3-6 hours
Systolic Pulmonary Artery Pressure (mmHg) | 3-6 hours
Right Atrium Pressure (mmHg) | 3-6 hours
  report measurement
Aortic Pulsatility Index (API) | 3-6 hours
  calculated measurement
Cardiac Power Input (W/m²) | 3-6 hours
Cardiac Power Output (Watts) | 3-6 hours
Stroke Volume (mL) | 3-6 hours
Cardiac Index (L/min/m²) | 3-6 hours
Cardiac Output (L/min) | 3-6 hours
Pulmonary Artery Oxygen Saturation (%) | 3-6 hours
Heart Rhythm | 3-6 hours
  Normal Sinus Rhythm, Atrial Fibrillation, Atrial Flutter, Ventricular Fibrillation, Ventricular Tachycardia, Sinus Bradycardia, Sinus Tachycardia, other
Heart Rate (beats per minute) | 3-6 hours
Mean Arterial Pressure (mmHg) | 3-6 hours
Diastolic Blood Pressure (mmHg) | 3-6 hours
Systolic Blood Pressure (mmHg) | 3-6 hours
Pulmonary Artery Compliance (mmHg) | 30 minutes
Right Ventricular Stroke Work Index (g·m-²·beat-¹) | 30 minutes
Pulmonary Artery Pulsatility Index (PAPi) | 30 minutes
  calculated measurement
Pulmonary Vascular Resistance (dynes/cm⁵) | 30 minutes
Systemic Vascular Resistance (mmHg/L/min) | 30 minutes
Pulmonary Capillary Wedge Pressure (mmHg) | 30 minutes
Diastolic Pulmonary Arterial Pressure (mmHg) | 30 minutes
Systolic Pulmonary Artery Pressure (mmHg) | 30 minutes
Right Atrium Pressure (mmHg) | 30 minutes
  report measurement
Aortic Pulsatility Index (API) | 30 minutes
  calculated measurement
Cardiac Power Input (W/m²) | 30 minutes
Stroke Volume (mL) | 30 minutes
Cardiac Power Output (Watts) | 30 minutes
Cardiac Index (L/min/m²) | 30 minutes
Cardiac Output (L/min) | 30 minutes
Pulmonary Artery Oxygen Saturation (%) | 30 minutes
Heart Rhythm | 30 minutes
  Normal Sinus Rhythm, Atrial Fibrillation, Atrial Flutter, Ventricular Fibrillation, Ventricular Tachycardia, Sinus Bradycardia, Sinus Tachycardia, other
Heart Rate (beats per minute) | 30 minutes
Mean Arterial Pressure (mmHg) | 30 minutes
Diastolic Blood Pressure (mmHg) | 30 minutes
Ultimate Disposition | Longitudinal Follow-Up (approximately 3 months)
  Heart recovery with discharge (alive)
Ultimate Disposition | Longitudinal Follow-Up (approximately 3 months)
  Left Ventricular Assist Device (LVAD)
Ultimate Disposition | Longitudinal Follow-Up (approximately 3 months)
  Transplant

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Delfiner, DO, MS, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No